CLINICAL TRIAL: NCT03729869
Title: Impact of Progesterone on Stress Reactivity and Cannabis Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aimee McRae-Clark, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00081360; 2U54DA016511-16 (NIH)
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Cannabis Use
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Progesterone Males (Experimental): 35 men will take 400 mg of progesterone a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Interventions: Drug: Progesterone
- Placebo Males (Placebo Comparator): 35 men will take placebo twice a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Interventions: Drug: Placebo
- Progesterone Female (Experimental): 35 women will take 200 mg of progesterone twice a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Interventions: Drug: Progesterone
- Placebo Females (Placebo Comparator): 35 women will take placebo twice a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — 200 mg of exogenous progesterone twice a day
  Other Names: Prometrium
  Arms: Progesterone Female; Progesterone Males
Drug: Placebo — One dose of matched placebo twice a day.
  Arms: Placebo Females; Placebo Males

SUMMARY:
This is a research study to find out if a hormone called progesterone affects marijuana users' stress response and marijuana use. Progesterone is a naturally occurring sex hormone involved in the menstrual cycle and reproduction, and has been shown to reduce withdrawal symptoms when people stop using substances like cocaine and nicotine. It is not FDA approved for treating cannabis users and is considered an investigational drug in this study.

DETAILED DESCRIPTION:
Participants will complete a screening visit to determine study eligibility. Eligible subjects will be scheduled to begin 22 days of study participation. During the first week, participants will be randomly assigned to take either progesterone or placebo (inactive medication) twice a day, and to abstain from marijuana use. During this week, participants will upload videos of themselves taking their medication and performing saliva drug tests. They will collect and store additional saliva samples each morning for hormone testing. They will also participate in "CREMA" sessions (Cue Reactivity Ecologic Momentary Assessment) three times a day. These sessions include looking at stressful and neutral pictures and rating stress and craving. At the end of this week, participants will return to the clinic and participate in a stress task. For the next two weeks, participants will continue to collect saliva samples and participate in CREMA sessions. They will return at the end of the two weeks to return study supplies. Urine samples will be collected at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.

  2. Meet DSM-5 criteria for moderate or severe cannabis use disorder (within the past three months) and report using cannabis at least five times weekly over the past month. While individuals may also meet criteria for mild use disorders of other substances, they must identify cannabis as their primary substance of abuse and must not meet criteria for any other moderate or severe substance use disorder (except tobacco) within the last 60 days.

  3. Age 18-45. 4. For women, regular menses (every 25-35 days). 5. Consent to remain abstinent from alcohol for 12 hours prior to study visits, and all other drugs other than cannabis or nicotine for the duration of the study.

  6. Women of childbearing potential must agree to utilize an effective means of birth control.

  7. Must consent to random assignment.

Exclusion Criteria:

* . Women who are pregnant, nursing or of childbearing potential and not practicing an effective means of birth control.

  2. Women who are amennorheic or using progesterone-based contraceptives. 3. Evidence or history of major medical illnesses, including liver diseases, abnormal vaginal bleeding, suspected or known malignancy, thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders, heart disease, diabetes, history of stroke or other medical conditions that the investigator deems as contraindicated for the individual to be in the study.

  4. History of or current psychotic disorder or bipolar affective disorder. 5. Current suicidal or homicidal ideation/risk. 6. Known allergy to progesterone or peanuts (vehicle for micronized progesterone).

  7. Unwilling or unable to maintain abstinence from alcohol 12 hours prior to study visits and all other drugs other than cannabis or nicotine for the duration of the study.

  8. Meet DSM-5 criteria for moderate or severe substance use disorder (other than nicotine or cannabis) within the past 60 days.

  9. Unable to comply with study procedures or pose threat to study staff.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone Males: 39 men will take 400 mg of progesterone a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Progesterone: 200 mg of exogenous progesterone twice a day
- Placebo Males: 41 men will take placebo twice a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Placebo: One dose of matched placebo twice a day.
- Placebo Females: 31 women will take placebo twice a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Placebo: One dose of matched placebo twice a day.
Period: Overall Study
Arm/Group | Progesterone Males | Placebo Males | Progesterone Female | Placebo Females
Started | 40 | 42 | 35 | 31
Completed | 39 | 41 | 35 | 31
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Progesterone Female: 34 women will take 200 mg of progesterone twice a day for 7 days and will complete a stress and marijuana cue reactivity task following the final dose.
  Progesterone: 200 mg of exogenous progesterone twice a day
- Total: Total of all reporting groups
Arm/Group | Progesterone Males | Placebo Males | Progesterone Female | Placebo Females | Total
Number analyzed (Participants) | 39 | 41 | 35 | 31 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 41 | 35 | 31 | 146
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 35 | 31 | 66
  Male | 39 | 41 | 0 | 0 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 6 | 5 | 10 | 8 | 29
  White | 32 | 35 | 24 | 23 | 114
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 35 | 31 | 146

OUTCOME MEASURES:

1. Primary Outcome: Cannabis Craving
Description: Subjects will rate marijuana craving on a 0-7 Likert scale where 0 is Not at All and 7 is extremely.
Time Frame: Immediately post stress/cue task.
Population: Males and females randomly assigned to take progesterone or placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Progesterone Males | Placebo Males | Progesterone Female | Placebo Females
Number analyzed (Participants) | 39 | 41 | 35 | 31
units on a scale | 3.7 (2.3) | 3.4 (2.2) | 4.3 (2.6) | 4.5 (2.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of study drug administration, Day 1, through follow-up on Day 21.
Arm/Group | Progesterone Males | Placebo Males | Progesterone Female | Placebo Females
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 0/35 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 26/39 | 28/41 | 24/35 | 23/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Progesterone Males (N=39) | Placebo Males (N=41) | Progesterone Female (N=35) | Placebo Females (N=31)
Headache (Nervous system disorders) | 9 (9) | 7 (7) | 9 (9) | 11 (11)
Marijuana withdrawal syndrome (General disorders) | 3 (3) | 8 (8) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 6 (6) | 4 (4) | 7 (7) | 4 (4)
Decreased appetite (Gastrointestinal disorders) | 8 (8) | 4 (4) | 6 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (4) | 9 (10) | 4 (4)
Hot Flush (Vascular disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Viral Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 6 (6) | 2 (2) | 8 (8)
Vivid Dreams/Nightmares (Psychiatric disorders) | 2 (2) | 1 (1) | 4 (5) | 4 (4)
Stomachache (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Mood swings (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Sleepiness (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Vaginal bleeding/spotting (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Abdominal cramps/discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Emotional lability (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT03729869/Prot_SAP_000.pdf